CLINICAL TRIAL: NCT00522717
Title: Enhancing Recovery After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Belinda Chen, Project Director, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 5R01NR009228-02 (NIH); R01NR009228 (NIH)
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease; Depression
MeSH Terms: conditions — Coronary Artery Disease; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- 2 (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — Subjects receive CBT in the home for 8 weeks with blood draws every other week during therapy.
  Arms: 1
Behavioral: Usual Care — Subjects receive Usual Care for 8 weeks followed by CBT
  Arms: 2

SUMMARY:
Patients recovering from coronary artery bypass graft (CABG) surgery have high rates of depression, and depression is associated with higher risk of complications and death. Recent discoveries show that depression involves changes in certain molecules in the blood, which are also involved in progressive coronary artery disease (CAD) and its complications. This study will evaluate the effects of cognitive behavioral therapy (CBT) as a treatment for depression on these biological markers among CABG patients.

ELIGIBILITY:
Inclusion Criteria:

* Undergone CABG at one of our recruitment sites

Exclusion Criteria:

* Less than 45 years of age
* Have cognitive impairment or major comorbid psychiatric conditions
* Have autoimmune disorder or malignancy
* Currently smoking

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Actual)
Dates: Start 2005-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Levels of proinflammatory cytokines (IL-1 and IL-6) | at baseline and after 8 weeks (at the completion of the intervention)
The soluble receptor for IL-6 (sIL-6) | at baseline and after 8 weeks (at the completion of the intervention)
Inflammatory markers c-reactive protein (CRP and sICAM-1) | at baseline and after 8 weeks (at the completion of the intervention)

SECONDARY OUTCOMES:
Depression symptoms (Beck Depression Inventory) | at baseline and after 8 weeks (at the completion of the intervention)
Presence of clinical depression | at baseline and after 8 weeks (at the completion of the intervention)
Pain | at baseline and after 8 weeks (at the completion of the intervention)
Sleep disturbances | at baseline and after 8 weeks (at the completion of the intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Doering, RN, DNSc, Principal Investigator — University of California, Los Angeles
Locations (5):
- United States (5):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente Medical Center - Sunset, Los Angeles, California
  - Department of Veterans Affairs-Greater Los Angeles Healthcare System, West Los Angeles, Los Angeles, California
  - University of California, Los Angeles School of Nursing, Los Angeles, California

REFERENCES:
- [Derived] Doering LV, Chen B, McGuire A, Bodan RC, Irwin MR. Persistent depressive symptoms and pain after cardiac surgery. Psychosom Med. 2014 Jul-Aug;76(6):437-44. doi: 10.1097/PSY.0000000000000074. PMID 24979578
- [Derived] Hwang B, Eastwood JA, McGuire A, Chen B, Cross-Bodan R, Doering LV. Cognitive behavioral therapy in depressed cardiac surgery patients: role of ejection fraction. J Cardiovasc Nurs. 2015 Jul-Aug;30(4):319-24. doi: 10.1097/JCN.0000000000000155. PMID 24763358